CLINICAL TRIAL: NCT01858740
Title: A Phase II Study of Selective Depletion of CD45RA+ T Cells From Allogeneic Peripheral Blood Stem Cell Grafts for the Prevention of GVHD in Children
Brief Title: Selective Depletion of CD45RA+ T Cells From Allogeneic Peripheral Blood Stem Cell Grafts in Preventing GVHD in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marie Bleakley, Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2660.00; NCI-2013-00958 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2660; 2660.00 (Other: Fred Hutch/University of Washington Cancer Consortium); K23CA154532 (NIH); RG9213077 (Other: Fred Hutch/University of Washington Cancer Consortium); R01HL121568 (NIH); 2P01CA018029 (NIH)
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Biphenotypic Leukemia; Acute Leukemia of Ambiguous Lineage; Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Myelodysplastic Syndrome With Excess Blasts-1; Myelodysplastic Syndrome With Excess Blasts-2; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Adult Acute Lymphoblastic Leukemia; Refractory Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — fludarabine phosphate; Methotrexate; merphos; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (CD45RA+ T cell depleted PBSCT) (Experimental): CONDITIONING REGIMEN: Patients undergo TBI BID on days -10 to -7, receive thiotepa IV over 4 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
  TRANSPLANT: Patients undergo CD34+ enriched, CD45RA+ T cell-depleted allogeneic PBSCT on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive tacrolimus IV continuously or PO every 12 hours beginning on day -1 and continuing through day 50 with taper. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Methotrexate; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo CD45RA+ T cell-depleted allogeneic peripheral blood stem cell transplant
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo CD45RA+ T cell-depleted allogeneic peripheral blood stem cell transplant
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation — Undergo CD45RA+ T cell-depleted allogeneic peripheral blood stem cell transplant
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well T cell depleted donor peripheral blood stem cell transplant works in preventing graft-versus-host disease in younger patients with high risk hematologic malignancies. Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Removing a subset of the T cells from the donor cells before transplant may stop this from happening.

DETAILED DESCRIPTION:
OUTLINE:

CONDITIONING REGIMEN: Patients undergo total body irradiation (TBI) twice daily (BID) on days -10 to -7, receive thiotepa intravenously (IV) over 4 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.

TRANSPLANT: Patients undergo CD34+ enriched, CD45RA+ T cell-depleted allogeneic PBSCT on day 0.

POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive tacrolimus IV continuously or orally (PO) every 12 hours beginning on day -1 and continuing through day 50 with taper. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed up for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are considered appropriate candidates for allogeneic hematopoietic stem cell transplantation and have one of the following diagnoses:

  * Acute lymphocytic leukemia in first or subsequent remission
  * Acute myeloid leukemia in first or subsequent remission
  * Acute lymphocytic leukemia in relapse or primary refractory disease with a circulating blast count of no more than 10,000/mm^3
  * Acute myeloid leukemia in relapse or primary refractory disease with a circulating blast count of no more than 10,000/mm^3
  * Refractory anemia with excess blasts (RAEB-1 and RAEB-2)
  * Chronic myelogenous leukemia with a history of accelerated phase or blast crisis
  * Other acute leukemia (including but not limited to 'biphenotypic', 'undifferentiated' or 'ambiguous lineage' acute leukemia)
* Patient with a human leukocyte antigen (HLA)-identical (HLA-A, B, C, and ribonucleic acid [RNA] binding motif protein 45 [DRB1] molecularly matched) unrelated donor or related donor capable of donating PBSC
* DONOR: HLA-matched unrelated donors (HLA-A, B, C, and DRB1 matched based on high-resolution typing) capable and willing to donate PBSC
* DONOR: HLA-matched related donors >= 18 years and capable and willing to donate PBSC

Exclusion Criteria:

* Patients with central nervous system (CNS) involvement refractory to intrathecal chemotherapy and/or standard cranial-spinal radiation
* Patients on other experimental protocols for prevention of acute GVHD
* Patients who weigh >= 70 kg must be discussed with the principal investigator prior to enrolling on the protocol
* Patients who are human immunodeficiency virus positive (HIV+)
* Patients with uncontrolled infections for whom myeloablative hematopoietic stem cell transplant (HCT) is considered contraindicated by the consulting infectious disease physician (upper respiratory tract viral infection does not constitute an uncontrolled infection in this context)
* Creatinine > 1.5 mg/dl
* Cardiac ejection fraction < 45%
* Patients who can perform pulmonary function tests will be excluded if they have a diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) of < 60% predicted; patients who are unable to perform pulmonary function tests (for example, due to young age and/or developmental status) will be excluded if the oxygen (O2) saturation is < 92% on room air
* Patients who have liver function test (LFTs) (including total bilirubin, aspartate aminotransferase [AST] and alanine aminotransferase [ALT]) >= twice the upper limit of normal should be evaluated by a gastrointestinal (GI) physician unless there is a clear precipitating factor (such as an azole, methotrexate, Bactrim or another drug); if the GI physician considers that HCT on protocol 2660 is contraindicated for that patient the patient will be excluded from the protocol; patients with Gilbert's syndrome and no other known liver function abnormality and patients with reversible drug-related transaminitis do not necessarily require GI consultation and may be included on the protocol
* Patients with a life expectancy < 3 months from co-existing disease other than the leukemia or RAEB
* Patients who are pregnant or breast-feeding
* Fertile patients of child bearing age unwilling to use contraception during and for 12 months post-transplant
* Patients with a significant other medical conditions that would make them unsuitable for transplant
* Patients with a known hypersensitivity to tacrolimus
* DONOR: Donors who are HIV-1, HIV-2, human T-lymphotropic virus (HTLV)-1, HTLV-2 seropositive or with active hepatitis B or hepatitis C virus infection
* DONOR: Donors who fail eligibility requirements for donation of cells or tissue per section 21 Code of Federal Regulations (CFR) 1271 for donation of a HCT/product (P) will be excluded unless use of the cells complies with 21 CFR 1271.65(b)(iii) (urgent medical need) or with 21 CFR 1271.65(b)(i) (allogeneic use in a first-degree or second-degree relative)
* DONOR: Unrelated donors donating outside of the United States of America (USA) or Germany

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bleakley, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Bleakley M, Sehgal A, Seropian S, Biernacki MA, Krakow EF, Dahlberg A, Persinger H, Hilzinger B, Martin PJ, Carpenter PA, Flowers ME, Voutsinas J, Gooley TA, Loeb K, Wood BL, Heimfeld S, Riddell SR, Shlomchik WD. Naive T-Cell Depletion to Prevent Chronic Graft-Versus-Host Disease. J Clin Oncol. 2022 Apr 10;40(11):1174-1185. doi: 10.1200/JCO.21.01755. Epub 2022 Jan 10. PMID 35007144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on referral for Hematopoietic Cell transplant at Fred Hutchinson Cancer Center between March 2014 and January 2017. The first participant was enrolled on April 10, 2014 and the last participant was enrolled on January 27, 2017.
Pre-assignment Details: Of the 20 patients enrolled, all 20 met inclusion criteria and went forward to be treated on the study.
Groups:
- Treatment (CD45RA+ T Cell Depleted PBSCT): CONDITIONING REGIMEN: Patients undergo TBI BID on days -10 to -7, receive thiotepa IV over 4 hours on days -6 and -5 and fludarabine phosphate IV over 30 minutes on days -6 to -2.
  TRANSPLANT: Patients undergo CD34+ enriched, CD45RA+ T cell-depleted allogeneic PBSCT on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive tacrolimus IV continuously or PO every 12 hours beginning on day -1 and continuing through day 50 with taper. Patients also receive methotrexate IV on days 1, 3, 6, and 11.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo CD45RA+ T cell-depleted allogeneic peripheral blood stem cell transplant
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Methotrexate: Given IV
  Peripheral Blood Stem Cell Transplantation: Undergo CD45RA+ T cell-depleted allogeneic peripheral blood stem cell transplant
  T Cell-Depleted Hematopoietic Stem Cell Transplantation: Undergo CD45RA+ T cell-depleted allogeneic peripheral blood stem cell transplant
  Tacrolimus: Given IV or PO
  Thiotepa: Given IV
  Total-Body Irradiation: Undergo TBI
Period: Overall Study
Arm/Group | Treatment (CD45RA+ T Cell Depleted PBSCT)
Started | 20
Day 28 Post Transplant | 20
Day 100 Post Transplant | 18
1 Year Post Transplant | 18
Completed | 16
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: All participants in single arm study received CD45RA+ T cell depletion PBSC transplant and IV Methotrexate and tacrolimus for GVHD prophylaxis (Day -1 to Day 50, then tapered from day 50)
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Graft Failure
Description: Graft failure defined as failure to reach ANC of >500/uL for 3 consecutive days by day 28, or irreversible decrease in ANC to <100 after an established donor graft. A reduction in ANC as result of relapse is not considered graft failure
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Participants: All participants in single arm study received CD45RA+ T cell depletion PBSC transplant and IV Methotrexate and tacrolimus for GVHD prophylaxis
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Participants
  Fail to engraft by D28 | 0
  Fail to maintain ANC >100 for 5 years | 1

2. Primary Outcome: Time to Discontinuation of Systemic Immunosuppression
Description: Measure the number of days to discontinuation of systemic immunosuppression (both including and excluding calcineurin inhibitors) in pediatric recipients of CD45RA+ T cell-depleted PBSCT. Possible outcomes range from no systemic immunosuppression (best outcome) to 5 years on immunosuppression (poor outcome)
Time Frame: 5 years post transplant
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Overall Study Patients Alive at D100: All participants in single arm study of CD45RA+ T cell depletion PBSC transplant and Methotrexate and tacrolimus for GVHD prophylaxis that were alive at D100
Arm/Group | Overall Study Patients Alive at D100
Number analyzed (Participants) | 18
Days
  Discontinuation (or never started) prednisone | 106 [87 to 238]
  Discontinuation of systemic immunosuppression (including calcineurin inhibitors) | 349 [266 to 405]

3. Secondary Outcome: Time to Platelet Count > 50,000/uL for 3 Days Without Transfusion
Description: Number of days post-transplant without transfusion where platelet count is >50,000/uL. Measured as the first of three days
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Days | 23 [21 to 29]

4. Secondary Outcome: Time to Platelet Count > 20,000/uL for 3 Days Without Transfusion
Description: Number of days post transplant until platelet count is >20,000/uL for three consecutive days without transfusion, counted as the first of three days
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Days | 19.5 [16 to 26]

5. Secondary Outcome: Time to ANC of > 1,000/uL
Description: Time (in days) to ANC of > 1,000/uL, counted as the first of three consecutive days post-transplant
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Days | 23 [19.75 to 28]

6. Secondary Outcome: Time to ANC of > 500/uL
Description: Time (in days) to ANC of > 500/uL, counted as the first of three consecutive days post-transplant
Time Frame: Up to 5 years
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Days | 20.5 [19 to 24]

7. Secondary Outcome: Occurrence of Chronic GHVD Meeting NIH Criteria and Requiring Systemic Pharmacological Immunosuppression
Description: Number of patients with chronic GVHD defined using NIH criteria. Incidents requiring only calcineurin inhibitors will not be counted. If patients do not develop cGVHD after transplant but then relapse and then receive a donor lymphocyte infusion or antigen specific T cells as treatment, they will no longer be evaluable for the cGVHD endpoint.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Patients Alive at D100
Number analyzed (Participants) | 18
Participants | 0

8. Secondary Outcome: Acute GVHD Grade III-IV
Description: Number of patients with acute GVHD grade III-IV
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Patients: All participants in single arm study received CD45RA+ T cell depletion PBSC transplant and IV Methotrexate and tacrolimus for GVHD prophylaxis
Arm/Group | Overall Study Patients
Number analyzed (Participants) | 20
Participants
  Grade III acute GVHD | 2
  Grade IV acute GVHD | 0

9. Secondary Outcome: Acute GVHD Grades II-IV
Description: Number of patients with acute GVHD grades II-IV
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Patients
Number analyzed (Participants) | 20
Participants
  Grade II acute GVHD | 15
  Grade III acute GVHD | 2
  Grade IV acute GVHD | 0

10. Secondary Outcome: Steroid Refractory Acute GVHD
Description: Presence of steroid refractory acute GVHD within the first 100 days post transplant
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Patients
Number analyzed (Participants) | 18
Participants | 0

11. Secondary Outcome: Relapse Post-transplant
Description: Relapse defined by the presence of malignant cells in marrow, peripheral blood, or extramedullary sites by histopathology
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Participants
  Relapse in first 100 days | 0
  Relapse between day 101 to 6 months | 0
  Relapse between 6 months to 1 year | 2
  Relapse between 1 to 5 years | 1
  Total relapse in first 5 years | 3

12. Secondary Outcome: Transplant Related Mortality
Description: Transplant related mortality defined as mortality in any patient for whom there has not been a diagnosis of relapse
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 20
Participants | 3

13. Secondary Outcome: Use of Additional Immune Suppressive Agents to Treat Chronic GVHD
Description: Use of additional immune suppressive agents to treat chronic GVHD other than first line therapy. First line therapy is considered prednisone and tacrolimus/cyclosporin.
Time Frame: Up to 5 years
Measure: Number; unit: Immunosuppressive agents
Arm/Group | Overall Study Patients Alive at D100
Number analyzed (Participants) | 18
Immunosuppressive agents | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs: Conditioning through D100; All cause mortality: Conditioning through 5 year
Groups:
- Treatment (CD45RA+ T Cell Depleted PBSCT): Single arm study: CD45RA+ T cell depletion PBSC transplant and Methotrexate and tacrolimus for GVHD prophylaxis (Day -1 to Day 50, then tapered from day 50)
Arm/Group | Treatment (CD45RA+ T Cell Depleted PBSCT)
All-Cause Mortality (participants affected / at risk) | 4/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (CD45RA+ T Cell Depleted PBSCT) (N=20)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (12)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 13 (15)
Vomiting (Gastrointestinal disorders) | 3 (3)
Multi-organ failure (General disorders) | 1 (1)
SOS/VOD (Hepatobiliary disorders) | 4 (4)
Enterocolitis infectious (Infections and infestations) | 1 (1)
C. difficile (Infections and infestations) | 3 (4)
CMV reactivation (Infections and infestations) | 6 (7)
Blood stream infections not including sepsis (Infections and infestations) | 8 (10)
Sepsis (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (10)
Aspartate aminotransferase increased (Investigations) | 2 (2)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 12 (12)
Neutrophil count decreased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 8 (8)
White blood cell decreased (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 10 (11)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (8)
Catheter related infection (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 3 (3)
Abdominal Infection (Infections and infestations) | 2 (2) — Colonic pneumatosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT01858740/Prot_SAP_000.pdf